CLINICAL TRIAL: NCT05690503
Title: Glutamatergic Modulation as a Treatment for Depressive Symptoms Among Patients With Post-acute Sequelae of COVID (PASC): A Pilot Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Elias Dakwar, Principal Investigator, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8336
Record Dates: First submitted 2022-12-30; First posted 2023-01-19 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Post-acute Sequelae of COVID-19; Depressive Symptoms; Cognitive Dysfunction
Keywords: Ketamine; PASC; Long Covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Depression; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CI-581a+CI-581b (Experimental): Administration of CI-581a at 0.8mg/kg during week 1. Administration of CI-581b at 0.025mg/kg during week 3.
  Interventions: Drug: CI-581a; Drug: CI-581b
- CI-581b+CI-581a (Experimental): Administration of CI-581b at 0.025mg/kg during week 1. Administration of CI-581a at 0.8mg/kg during week 3.
  Interventions: Drug: CI-581a; Drug: CI-581b

INTERVENTIONS:
Drug: CI-581a — Medication infusion intravenously over 90 minutes.
Drug: CI-581b — Medication infusion intravenously over 90 minutes.

SUMMARY:
Post-acute sequelae of SARS-CoV2 (PASC), colloquially known as "long-COVID," is thought to affect between 10-30% of all COVID-19 survivors. Patients with PASC also report worsening behavioral health symptoms over time that include new-onset depression, anxiety, and even suicidal behavior. The purpose of this randomized, double-blind, controlled trial is to test the efficacy of a glutamate modulator among PASC patients suffering from new-onset or worsening of depressive symptoms.

DETAILED DESCRIPTION:
While PASC symptoms have been identified in nearly every organ system, the most common symptoms include fatigue, cognitive and attention deficits (known as 'brain fog'), shortness of breath, and post-exertional malaise. New-onset depression, anxiety, and even suicidal behavior have also been reported. Symptoms of PASC can exhibit daily variation; additionally PASC frequently demonstrates a relapsing and remitting course. This is mitigated by cognitive and emotional stress, physical exertion, diet, and alcohol consumption; therefore, measuring treatment response and the course of illness over time can be challenging. While there are many ongoing trials evaluating a variety of treatments for PASC, no clear treatment has emerged; additionally, there are no published data on psychotropic medications alleviating the inflammatory response and psychiatric symptoms in PASC.

Alterations in the transmission between neurons of a neurotransmitter called glutamate are an important target of pharmacotherapy for PASC. Glutamate modulators have demonstrated promise in improving depressive symptoms and suicidality and can improve cognitive functioning among patients with these symptoms. The study team has recently developed a novel design that integrates a clinical trial involving serial infusions. The current trial will evaluate the effect of a sub-anesthetic infusion on individuals with PASC and depressive symptoms who complete a randomized, double-blind, placebo-controlled pilot study conducted over 5 weeks using a cross-over and counterbalanced design.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the case-definition for PASC with depressive symptoms
2. Otherwise physically healthy
3. No adverse reactions to study medications
4. Capacity to consent and comply with study procedures, including sufficient proficiency in English
5. Sexually active participants must use an effective form of birth control (condom plus spermicide, diaphragm plus spermicide, or birth control pills) before and throughout their study participation.
6. Willingness to provide one or more emergency contacts to the study team

Exclusion Criteria:

1. Meeting the DSM-5 criteria for lifetime history of bipolar disorder, schizophrenia, or any psychotic illness.
2. Lifetime history of delirium, dementia, amnesia, or dissociative disorders
3. Current suicide risk or a history of suicide attempt within the past year
4. Pregnant or interested in becoming pregnant during the study period.
5. Any of the following cardiac conditions: clinically significant left ventricular hypertrophy, angina, clinically significant arrhythmia within 1 year of signing study consent form.
6. Unstable physical disorders which might make participation hazardous such as hypertension (>160/90), anemia, active hepatitis or other liver disease (transaminase levels <3 X the upper limit of normal will be considered acceptable), epilepsy, or untreated diabetes. Participants reporting HIV+ status will be asked to provide information about their current treatment, including all medications. Participants who are on the antiretroviral ritonavir (Norvir) will be excluded due to the possibility that ketamine in combination with this medication may increase the risk of drug-induced hepatitis.
7. Previous history of a substance use disorder with the study medications, and/or a history of an adverse reaction/experience with prior exposure to the study medications.
8. Recent history of significant violence (past 2 years) leading to an individual incurring physical harm, police involvement, or resulting in legal action.
9. On psychotropic or other medications whose effect could be disrupted by participation in the study.
10. Other personal circumstances and behavior judged to be incompatible with establishment of rapport or safe exposure to the study medications.
11. Physiologic dependence on a substance including benzodiazepines, alcohol, or opioids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in depressive symptoms | from baseline to week 5.

SECONDARY OUTCOMES:
Improvement in neurocognitive symptoms of PASC | from baseline to week 5.

CONTACTS AND LOCATIONS:
Overall Officials: Saleena Subaiya, MD, Principal Investigator — New York State Psychiatric Institute; Elias Dakwar, MD, Principal Investigator — New York State Psychiatric Institute; Kate O'Malley, MA, Study Director — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States